CLINICAL TRIAL: NCT06082323
Title: A Phase 1，Randomized, Placebo-controlled, Single and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered LT-002-158 in Healthy Adult Volunteers
Brief Title: A Single and Multiple Ascending Dose Trial of LT-002-158 Tablets in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Leadingtac Pharmaceutical (Shaoxing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT2158CHN001V6
Record Dates: First submitted 2023-09-26; First posted 2023-10-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteer; Hidradenitis Suppurativa; Atopic Dermatitis
MeSH Terms: conditions — Hidradenitis Suppurativa; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single Ascending Dose (SAD) (Experimental): Part 1: healthy volunteer subject cohorts randomized 6:2 receiving a single dose of LT-002-158 or placebo. The first cohort will receive 50mg of LT-002-158 or placebo. Dose escalation will occur if LT-002-158 or placebo is tolerated.
  Interventions: Drug: LT-002-158/Placebo oral tablet(s)
- Food effect (Experimental): Part 2: A 3-treatment, 3 period crossover study will be conducted, which is composed of 15 healthy Volunteer subjects, who will be receiving a single dose of LT-002-158 in fasted, standard meal and high fat meal.
  Interventions: Drug: LT-002-158/Placebo oral tablet(s)
- Multiple Ascending Doses (MAD) Study (Experimental): Part 3: Healthy volunteer subject cohorts randomized 8:2 to receive LT-002-158 or placebo for 14 days continuous dosing. The first cohort will receive a dose of LT-002-15 or placebo determined to be safe based on data generated in the SAD portion and FE study.
  Interventions: Drug: LT-002-158/Placebo oral tablet(s)

INTERVENTIONS:
Drug: LT-002-158/Placebo oral tablet(s) — Single ascending dose escalation and multiple ascending dose escalation study followed by an evaluation of food effects on absorption Masking: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
  Other Names: LT-002-158

SUMMARY:
LT-002-158 is an oral IRAK4 protein degrader being developed for the treatment of autoimmune disease and inflammation including Hidradenitis Suppurativa and Atopic Dermatitis. This first-in-human (FIH) study will characterize the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of a single ascending dose and multiple ascending doses of LT-002-158 in healthy volunteers. The effects of food on the pharmacokinetics of LT-002-158 will also be assessed in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1 randomized, placebo-controlled, single and multiple ascending dose trial of LT-002-158 that will characterize the safety, PK and PD of orally administered LT-002-158 after a single dose (Part 1) and after repeated dosing in healthy adult volunteers (Part 3). A 3 treatment, 3-periods crossover design is planned on healthy subjects to understand food effects (FE) on the PK of LT-002-158 (Part 2). Once adequate safety and PK data from multiple SAD cohorts and FE cohort become available, a safe starting dose for the 14-day MAD portion of the study will be selected so as to initiate the enrolment of healthy subjects into 14-day multiple ascending dose (MAD) escalation cohorts.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy volunteers who fully understand the content, process, and possible adverse event of the study and capable of giving written informed consent form.

  2) Male or female between 18 and 55 years of age (inclusive), at the time of signing the informed consent form.

  3) Body mass index (BMI) range within 18~30 kg/m2 (inclusive), and body weight of ≥ 50.0 kg for male and ≥ 45.0 kg for female.

  4) Healthy volunteers who must be confirmed as negative in the SARS-CoV-2 test on Day -2 (admission).

  5) Healthy volunteers with no significant medical history judged by the Investigator and in good health, fully physical examinations, vital signs, 12-lead electrocardiograms (12-ECGs), clinical laboratory tests (hematology, urinalysis, blood chemistry and coagulation test), serum virology test.

  6) Females must be non- pregnant, non- lactating and must have negative serum pregnancy test at screening. Women of child bearing potential and males must be willing to use highly effective acceptable forms of contraception from screening to 6 months after the last study drug administration. Males and females must be willing to avoid donating sperm or egg respectively during the study period and 6 months after the last dose of IP.

  7) All HVs who must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Healthy volunteers with history of allergy, including anaphylaxis to food, drugs, or are allergic to any component of the IP considered clinically significant in the Investigator's judgment.
2. Healthy volunteers who are vegans or have medical dietary restrictions.
3. Healthy volunteers with clinically relevant history of respiratory, immunological, dermatological, connective tissue, lymphatic, metabolism, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, urinary, endocrine, neurologic disorders, psychiatric, and/ or any other conditions, judged by the Investigator, that would make the healthy volunteer unsuitable for this study.
4. Healthy volunteers who have acute GI symptoms at screening or admission (e.g., nausea, vomiting, diarrhea, heartburn).
5. Healthy volunteers who have an acute infection such as influenza at screening or admission.
6. Healthy volunteers who have increased risk of infection.

   1. With history and/or presence of tuberculosis; positive result for IFN-γ release assay (IGRA) (i.e., QuantiFERON TB-Gold), the test may be repeated if the initial test result is indeterminate. Volunteers who have resided in regions where tuberculosis or mycosis are endemic during 90 days before screening or who intend to visit such a region during the duration of the study.
   2. HV who engage in high risk unsafe sexual practices.
   3. With active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
   4. With a disease history suggesting abnormal immune function.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of LT-002-158 following single dose in HVs | up to 28 days
  Incidence and severity of treatment emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chen, MD, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Distric Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldburg SR, Strober BE, Payette MJ. Hidradenitis suppurativa: Epidemiology, clinical presentation, and pathogenesis. J Am Acad Dermatol. 2020 May;82(5):1045-1058. doi: 10.1016/j.jaad.2019.08.090. Epub 2019 Oct 9. PMID 31604104